CLINICAL TRIAL: NCT06380062
Title: Pre-operative Plasma Concentrations of Choline and Its Metabolites in People With Prostate Cancer Compared to Those With Benign Hyperplasia
Brief Title: Choline Metabolites in People With Prostate Cancer and Those With Benign Hyperplasia
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Rima Obeid, Prof. Dr., Universität des Saarlandes
Other Study IDs: Choline Prostate Cancer
Record Dates: First submitted 2023-05-02; First posted 2024-04-23 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Primary Prostate Urothelial Cancer; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary prostate cancer: Men participants diagnosed with primary prostate cancer are "cases"
  Interventions: Other: Plasma concentration of choline
- Benign hyperplasia: Men participants diagnosed with benign hyperplasia are the "controls"
  Interventions: Other: Plasma concentration of choline

INTERVENTIONS:
Other: Plasma concentration of choline — The exposure in this observational study is plasma concentrations of choline

SUMMARY:
The aim of this study was to investigate plasma concentrations of one-carbon metabolites and phospholipid classes in participants with primary prostate cancer and those with benign hyperplasia. Moreover, the metabolites were studied in relation to tumor grade and age.

DETAILED DESCRIPTION:
This observational study recruited participants with primary prostate cancer (cases) and those with benign hyperplasia (controls) before the surgery. Data on the outcomes of the surgery including the results of the biopsy investigation were collected. Blood samples were collected before the surgery in context of routine blood investigations. Blood plasma samples collected on ethylenediaminetetraacetic acid (EDTA) were used to measure concentrations of free choline, betaine, dimethylglycine, folate forms, S-adenosylhomocysteine, S-adenosylmethionine, homocysteine, cystathionine, and methylmalonic acid (MMA). Data on serum concentrations of prostate specific antigen (PSA) and the tumor grade and classification (Gleason Score system) were collected. The associations between the plasma concentrations of the metabolites and PSA or the Gleason score were studied. The concentrations of the metabolic markers were compared between the cases and the controls according to the age of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Men participants
* age > 50 years
* recently diagnosed with primary prostate cancer or benign hyperplasia

Exclusion Criteria:

* vitamin B supplementation (folic acid> 400 µg / day; B12> 10 µg / day; B6> 10 mg / day)
* renal failure
* advanced liver disease
* chronic alcohol consumption
* metastases
* methotrexate therapy.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with prostate cancer or benign hyperplasia
Study Population: Participants were recruited before carrying out the radical prostatectomy surgery, or TURP surgery.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2012-01-12 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Plasma choline concentrations | through study completion, on average 1 year
  Concentrations measured in plasma with liquid chromatography tandem mass spectrometry
Whole blood choline concentrations | through study completion, on average 1 year
  Concentrations measured in plasma with liquid chromatography tandem mass spectrometry

SECONDARY OUTCOMES:
Plasma and whole blood folate forms | through study completion, on average 1 year
  Concentrations measured in plasma with liquid chromatography tandem mass spectrometry
Plasma phospholipids | through study completion, on average 1 year
  Concentrations measured in plasma with liquid chromatography tandem mass spectrometry after extraction
Plasma S-adenosylmethionine concentrations | through study completion, on average 1 year
  Concentrations measured in plasma with liquid chromatography tandem mass spectrometry
Plasma betaine concentrations | through study completion, on average 1 year
  Concentrations measured in plasma with liquid chromatography tandem mass spectrometry
Plasma methylmalonic acid concentrations | through study completion, on average 1 year
  Concentrations measured in plasma with gas chromatography mass spectrometry
Plasma homocysteine concentrations | through study completion, on average 1 year
  Concentrations measured in plasma with liquid chromatography tandem mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Rima Obeid, PhD, Principal Investigator — Saarland University Hospital
Locations (1):
- University of Saarland, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. Only data in aggregated form can be provided upon reasonable request to the study PI.

REFERENCES:
- [Result] Awwad HM, Ohlmann CH, Stoeckle M, Aziz R, Geisel J, Obeid R. Choline-phospholipids inter-conversion is altered in elderly patients with prostate cancer. Biochimie. 2016 Jul;126:108-14. doi: 10.1016/j.biochi.2016.01.003. Epub 2016 Jan 14. PMID 26776756
- [Result] Awwad HM, Ohlmann CH, Stoeckle M, Geisel J, Obeid R. Serum concentrations of folate vitamers in patients with a newly diagnosed prostate cancer or hyperplasia. Clin Biochem. 2018 Jun;56:41-46. doi: 10.1016/j.clinbiochem.2018.04.011. Epub 2018 Apr 16. PMID 29673813